CLINICAL TRIAL: NCT03505099
Title: A Global Study of a Single, One-Time Dose of AVXS-101 Delivered to Infants With Genetically Diagnosed and Pre-symptomatic Spinal Muscular Atrophy With Multiple Copies of SMN2
Brief Title: Pre-Symptomatic Study of Intravenous Onasemnogene Abeparvovec-xioi in Spinal Muscular Atrophy (SMA) for Patients With Multiple Copies of SMN2
Acronym: SPR1NT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Gene Therapies (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVXS-101-CL-304; 2017-004087-35 (EudraCT Number); JapicCTI-184203 (Registry Identifier: JapicCTI); COAV101A12303 (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Spinal Muscular Atrophy
Keywords: gene therapy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Zolgensma

STUDY DESIGN:
Intervention Model Description: Open-label, single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- onasemnogene abeparvovec-xioi (Experimental): One-time intravenous infusion of onasemnogene abeparvovec-xioi at 1.1 X 10^14 vg/kg
  Interventions: Biological: onasemnogene abeparvovec-xioi

INTERVENTIONS:
Biological: onasemnogene abeparvovec-xioi — A non-replicating recombinant AAV9 containing the complimentary deoxyribonucleic acid (cDNA) of the human SMN gene under the control of the cytomegalovirus (CMV) enhancer/chicken-β-actin-hybrid promoter (CB). The AAV inverted terminal repeat (ITR) has been modified to promote intramolecular annealing of the transgene, thus forming a double-stranded transgene ready for transcription.
  Other Names: Zolgensma

SUMMARY:
To evaluate the safety and efficacy of intravenous onasemnogene abeparvovec-xioi in pre-symptomatic patients with SMA and 2 or 3 copies SMN2

DETAILED DESCRIPTION:
Phase 3, open-label, single-arm study of a single, one-time dose of onasemnogene abeparvovec-xioi (gene replacement therapy) in patients with spinal muscular atrophy who meet enrollment criteria and are genetically defined by bi-allelic deletion of survival motor neuron 1 gene (SMN1) with 2 or 3 copies of survival motor neuron 2 gene (SMN2). Patients with SMN1 point mutations or the SMN2 gene modifier mutation (c.859G>C) may enroll but will not be included in the efficacy analysis sets.

The study includes a screening period, a gene replacement therapy period, and a follow-up period. During the screening period (Days -30 to -2), patients whose parent(s)/legal guardian(s) provide informed consent will undergo screening procedures to determine eligibility for study enrollment. Patients who meet the entry criteria will enter the in-patient gene replacement therapy period (Day -1 to Day 2). On Day -1, patients will be admitted to the hospital for pre-treatment baseline procedures. On Day 1, patients will receive a single, one-time intravenous (IV) infusion of onasemnogene abeparvovec-xioi, and will undergo in-patient safety monitoring for a minimum of 24 hours post infusion. Patients may be discharged 24 hours (48 hours in Japan) after the infusion, based on Investigator judgment. During the outpatient follow-up period (Days 3 to End of Study at 18 or 24 of age, dependent upon respective SMN2 copy number), patients will return at regularly scheduled intervals for efficacy and safety assessments until the End of Study when the patient reaches 18 months of age (SMN2 = 2) or 24 months of age (SMN2 = 3). After the End of Study visit, eligible patients will be invited to rollover into a long-term follow up study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤6 weeks (≤42 days) at time of dose
* Ability to tolerate thin liquids as demonstrated through a formal bedside swallowing test
* Compound muscle action potential (CMAP) ≥2mV at Baseline; centralized review of CMAP data will be conducted
* Gestational age of 35 to 42 weeks
* Parent(s)/legal guardian(s) willing and able to complete the informed consent process and comply with study procedures and visit schedule

  * Patients with pre-symptomatic SMA Type 1 as determined by the following features:

    a. 2 copies of SMN2 (n ≥14)
  * Patients with pre-symptomatic SMA Type 2 as determined by the following features:

    1. 3 copies of SMN2 (n ≥12)

Exclusion Criteria:

* Weight at screening visit <2 kg
* Hypoxemia (oxygen saturation <96% awake or asleep without any supplemental oxygen or respiratory support) at the screening visit or for altitudes >1000 m, oxygen saturation <92% awake or asleep without any supplemental oxygen or respiratory support at the screening visit
* Any clinical signs or symptoms at screening or immediately prior to dosing that are, in the opinion of the Investigator, strongly suggestive of SMA
* Tracheostomy or current prophylactic use or requirement of noninvasive ventilatory support at any time and for any duration prior to screening or during the screening period
* Patients with signs of aspiration/inability to tolerate nonthickened liquids based on a formal swallowing test performed as part of screening or patients receiving any non-oral feeding method
* Clinically significant abnormal laboratory values (gamma-glutamyl transferase [GGT], Alanine transaminase [ALT], and aspartate aminotransferase [AST], or total bilirubin > 2 × the upper limit of normal [ULN], creatinine ≥ 1.0 mg/dL, hemoglobin [Hgb] < 8 or > 18 g/dL; white blood cell [WBC] > 20,000 per cmm) prior to gene replacement therapy. Patients with an elevated bilirubin level that is unequivocally the result of neonatal jaundice shall not be excluded
* Treatment with an investigational or commercial product, including nusinersen, given for the treatment of SMA. This includes any history of gene therapy, prior antisense oligonucleotide treatment, or cell transplantation.
* Patients whose weight-for-age is below the third percentile based on World Health Organization (WHO) Child Growth Standards
* Biological mother with active viral infection as determined by screening laboratory samples (includes human immunodeficiency virus [HIV] or positive serology for hepatitis B or C)

  • Biological mothers with clinical suspicion of Zika virus that meet Centers for Disease Control and Prevention (CDC) Zika virus epidemiological criteria including history of residence in or travel to a geographic region with active Zika transmission at the time of travel will be tested for Zika virus RNA. Positive results warrant confirmed negative Zika virus RNA testing in the patient prior to enrollment.
* Serious nonrespiratory tract illness requiring systemic treatment and/or hospitalization within 2 Weeks prior to screening
* Upper or lower respiratory infection requiring medical attention, medical intervention, or increase in supportive care of any manner within 4 Weeks prior to dosing
* Severe nonpulmonary/respiratory tract infection within 4 Weeks before administration of gene replacement therapy or concomitant illness that, in the opinion of the Investigator or Sponsor medical monitor, creates unnecessary risks for gene replacement therapy such as:

  * Major renal or hepatic impairment
  * Known seizure disorder
  * Diabetes mellitus
  * Idiopathic hypocalciuria
  * Symptomatic cardiomyopathy
* Known allergy or hypersensitivity to prednisolone or other glucocorticosteroids or their excipients
* Previous, planned or expected major surgical procedure including scoliosis repair surgery/procedure during the study assessment period
* Concomitant use of any of the following: drugs for treatment of myopathy or neuropathy, agents used to treat diabetes mellitus, or ongoing immunosuppressive therapy, plasmapheresis, immunomodulators such as adalimumab, immunosuppressive therapy within 4 Weeks prior to gene replacement therapy
* AntiAAV9 antibody titer >1:50 as determined by Enzyme-linked Immunosorbent Assay (ELISA) binding immunoassay

  • Should a potential patient demonstrate AntiAAV9 antibody titer >1:50, he or she may receive retesting inside the 30-Day screening period and will be eligible to participate if the AntiAAV9 antibody titer upon retesting is ≤1:50, provided the <6 Week age requirement at the time of dosing is still met
* Biological mother involved with the care of the child refuses anti-AAV9 antibody testing prior to dosing

Max Age: 42 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (11):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Hospital, Orlando, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Clinic for Special Children, Strasburg, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - University Hospital and UW Health Clinics, Madison, Wisconsin
- Sydney Children's Hospital, Randwick, New South Wales, Australia
- Centre Hospitalier Régional Hôpital La Citadelle, Liège, Belgium
- Canada Childrens Hospital of Eastern Ontario, Ottawa, Ontario, Canada
- Tokyo Women's Medical, Tokyo, Japan
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Strauss KA, Farrar MA, Muntoni F, Saito K, Mendell JR, Servais L, McMillan HJ, Finkel RS, Swoboda KJ, Kwon JM, Zaidman CM, Chiriboga CA, Iannaccone ST, Krueger JM, Parsons JA, Shieh PB, Kavanagh S, Wigderson M, Tauscher-Wisniewski S, McGill BE, Macek TA. Onasemnogene abeparvovec for presymptomatic infants with three copies of SMN2 at risk for spinal muscular atrophy: the Phase III SPR1NT trial. Nat Med. 2022 Jul;28(7):1390-1397. doi: 10.1038/s41591-022-01867-3. Epub 2022 Jun 17. PMID 35715567
- [Derived] Strauss KA, Farrar MA, Muntoni F, Saito K, Mendell JR, Servais L, McMillan HJ, Finkel RS, Swoboda KJ, Kwon JM, Zaidman CM, Chiriboga CA, Iannaccone ST, Krueger JM, Parsons JA, Shieh PB, Kavanagh S, Tauscher-Wisniewski S, McGill BE, Macek TA. Onasemnogene abeparvovec for presymptomatic infants with two copies of SMN2 at risk for spinal muscular atrophy type 1: the Phase III SPR1NT trial. Nat Med. 2022 Jul;28(7):1381-1389. doi: 10.1038/s41591-022-01866-4. Epub 2022 Jun 17. PMID 35715566
- [Derived] Day JW, Mendell JR, Mercuri E, Finkel RS, Strauss KA, Kleyn A, Tauscher-Wisniewski S, Tukov FF, Reyna SP, Chand DH. Clinical Trial and Postmarketing Safety of Onasemnogene Abeparvovec Therapy. Drug Saf. 2021 Oct;44(10):1109-1119. doi: 10.1007/s40264-021-01107-6. Epub 2021 Aug 12. PMID 34383289
- See also: Novartis Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17902
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 participants took part in the trial at 16 sites in the United States, the United Kingdom, Belgium, Canada, Australia and Japan between April 2018 and June 2021.
Pre-assignment Details: A total of 44 participants were screened, of which 14 were screen failures and 30 were enrolled and received study drug. One participant had 4 copies of SMN2. This participant was excluded from all analysis populations and data is not reported due to privacy concerns.
Groups:
- Cohort 1: Bi-allelic Deletions of SMN1 and 2 Copies of SMN2: Participants with bi-allelic deletions of survival of motor neuron 1 (SMN1) and 2 copies of SMN2 received a single dose of AVXS-101 administered as an intravenous (IV) infusion over 60 minutes at a dose of 1.1 × 10^14 vg/kg (vector genome per kilogram) on Day 1 of the overall study. Participants also received daily doses of prophylactic oral prednisolone starting at a dose of 1-2 mg/kg/day from 1 day prior to AVXS-101 infusion until at least 30 days post-infusion at which point the prednisolone dose could be tapered downwards. At week 9, prednisolone could be discontinued.
- Cohort 2: Bi-allelic Deletions of SMN1 and 3 Copies of SMN2: Participants with bi-allelic deletions of SMN1 and 3 copies of SMN2 received a single dose of AVXS-101 administered as an IV infusion over 60 minutes at a dose of 1.1 × 10^14 vg/kg on Day 1 of the overall study. Participants also received daily doses of prophylactic oral prednisolone starting at a dose of 1-2 mg/kg/day from 1 day prior to AVXS-101 infusion until at least 30 days post-infusion at which point the prednisolone dose could be tapered downwards. At week 9, prednisolone could be discontinued.
Period: Overall Study
Arm/Group | Cohort 1: Bi-allelic Deletions of SMN1 and 2 Copies of SMN2 | Cohort 2: Bi-allelic Deletions of SMN1 and 3 Copies of SMN2
Started | 14 | 15
Received AVXS-101 | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Bi-allelic Deletions of SMN1 and 2 Copies of SMN2 | Cohort 2: Bi-allelic Deletions of SMN1 and 3 Copies of SMN2 | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 15 | 29
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 2 | 4
  American Indian or Alaska Native | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 7 | 10 | 17
  Other | 4 | 2 | 6
SMN2 gene modifier mutation (c.859G>C) Present [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Number of Participants Who Achieved Sitting Alone for at Least 30 Seconds
Description: Defined by the Bayley Scales of Infant and Toddler Development (BSID) Gross Motor (GM) subtest performance criteria number 26, confirmed by video recording, as a participant who sits for at least 30 seconds without assistance from another person or object. The participant was allowed to use their upper extremities.
Time Frame: From Day 1 up to 18 months of age visit
Population: Intent-to-Treat (ITT) population (cohort 1) - All enrolled participants with bi-allelic SMN1 deletions and 2 copies of SMN2 without the SMN2 gene modifier mutation (c.859G>C) who received AVXS-101.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Bi-allelic Deletions of SMN1 and 2 Copies of SMN2
Number analyzed (Participants) | 14
Participants | 14

2. Primary Outcome: Cohort 2: Number of Participants Who Achieved Standing Alone for at Least 3 Seconds
Description: Defined by the BSID GM subtest performance criteria number 40, confirmed by video recording, as a participant who stands alone for at least 3 seconds unsupported.
Time Frame: From Day 1 up to 24 months of age visit
Population: ITT population (cohort 2) - All enrolled participants with bi-allelic SMN1 deletions and 3 copies of SMN2 without the SMN2 gene modifier mutation (c.859G>C) who received AVXS-101.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Bi-allelic Deletions of SMN1 and 3 Copies of SMN2
Number analyzed (Participants) | 15
Participants | 15
Statistical Analysis 1: Comparison: Cohort 2: Bi-allelic Deletions of SMN1 and 3 Copies of SMN2; Test type: Superiority; p < 0.0001, Fisher Exact; Difference of Proportion = 76.5, 95% CI 2-sided [50.95 to 92.21]; Data for the current study were compared to historical control data (Finkel et al, 2014 - PubMed 25080519) where 19 out of 81 participants (23.46%) with 3 copies of SMN2 achieved standing alone for at least 3 seconds

3. Secondary Outcome: Cohort 1: Event-free Survival at 14 Months of Age
Description: Event-free survival at 14 months of age was defined as the number of participants who did not die, did not require permanent ventilation and did not withdraw from the study by 14 months of age.
Time Frame: From Day 1 up to 14 months of age
Population: ITT population (cohort 1) - All enrolled participants with bi-allelic SMN1 deletions and 2 copies of SMN2 without the SMN2 gene modifier mutation (c.859G>C) who received AVXS-101.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Bi-allelic Deletions of SMN1 and 2 Copies of SMN2
Number analyzed (Participants) | 14
Participants | 14
Statistical Analysis 1: Comparison: Cohort 1: Bi-allelic Deletions of SMN1 and 2 Copies of SMN2; Test type: Superiority; p < 0.0001, Fisher Exact; Difference of Proportion = 73.9, 95% CI 2-sided [44.67 to 91.61]; Data for the current study were compared to historical control data (Finkel et al 2014 - PubMed 25080519) where 6 out of 23 participants (26.09%) with 2 copies of SMN2 were alive and did not require permanent ventilation

4. Secondary Outcome: Cohort 1: Number of Participants Who Achieved the Ability to Maintain Weight at or Above the Third Percentile Without the Need for Non-Oral or Mechanical Feeding Support
Description: The ability to maintain weight at or above the third percentile without the need for non-oral or mechanical feeding support was defined by meeting the following criteria at each visit up to 18 months of age:
  * Did not receive nutrition through mechanical support (i.e., feeding tube)
  * Maintained weight (≥ third percentile for age and sex as defined by World Health Organization [WHO] guidelines) consistent with the participant's age at the assessment.
Time Frame: From Day 1 up to 18 months of age
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Bi-allelic Deletions of SMN1 and 2 Copies of SMN2
Number analyzed (Participants) | 14
Participants | 13

5. Secondary Outcome: Cohort 2: Number of Participants Who Achieved the Ability to Walk Alone
Description: Defined by the BSID GM subtest performance criteria number 43, confirmed by video recording, as a participant who takes 5 coordinated independent steps.
Time Frame: From Day 1 up to 24 months of age visit
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Bi-allelic Deletions of SMN1 and 3 Copies of SMN2
Number analyzed (Participants) | 15
Participants | 14
Statistical Analysis 1: Comparison: Cohort 2: Bi-allelic Deletions of SMN1 and 3 Copies of SMN2; Test type: Superiority; p < 0.0001, Fisher Exact; Difference of Proportion = 72.3, 95% CI 2-sided [44.90 to 90.11]; Data for the current study were compared to historical control data (Finkel et al, 2014 - PubMed 25080519) where 17 out of 81 participants (20.99%) with 3 copies of SMN2 achieved the ability to walk alone

ADVERSE EVENTS:
Time Frame: Cohort 1: Treatment-emergent adverse events (TEAEs) were collected from Day 1 up to the 18 months of age visit. Serious adverse events (SAEs) were collected from signing of informed consent to 30 days after the last study visit (up to a maximum of approximately 20 months). Cohort 2: TEAEs were collected from Day 1 up to the 24 months of age visit. SAEs were collected from signing of informed consent to 30 days after the last study visit (up to a maximum of approximately 26 months).
Arm/Group | Cohort 1: Bi-allelic Deletions of SMN1 and 2 Copies of SMN2 | Cohort 2: Bi-allelic Deletions of SMN1 and 3 Copies of SMN2
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 5/14 | 3/15
Other Adverse Events (participants affected / at risk) | 14/14 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Bi-allelic Deletions of SMN1 and 2 Copies of SMN2 (N=14) | Cohort 2: Bi-allelic Deletions of SMN1 and 3 Copies of SMN2 (N=15)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Bi-allelic Deletions of SMN1 and 2 Copies of SMN2 (N=14) | Cohort 2: Bi-allelic Deletions of SMN1 and 3 Copies of SMN2 (N=15)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Precocious puberty (Endocrine disorders) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 3 (4)
Gingival pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 2 (2) | 5 (6)
Tooth development disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Developmental delay (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 11 (18)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Candida nappy rash (Infections and infestations) | 1 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (2) | 1 (2)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 2 (3) | 1 (3)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 3 (4)
Otitis media (Infections and infestations) | 1 (1) | 3 (6)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (2)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Rhinovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 9 (13)
Viral upper respiratory tract infection (Infections and infestations) | 3 (10) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Exanthema subitum (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (3)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 2 (2)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Roseola (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheal deviation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 4 (6)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1)
Head lag (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 1 (2) | 2 (2)
Bacterial test positive (Investigations) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 0 (0) | 2 (2)
Carbon dioxide decreased (Investigations) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Poor feeding infant (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hip deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Areflexia (Nervous system disorders) | 2 (2) | 1 (2)
Hypertonia (Nervous system disorders) | 1 (1) | 0 (0)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0)
Hyporeflexia (Nervous system disorders) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 3 (5) | 2 (3)
Motor developmental delay (Nervous system disorders) | 1 (1) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 3 (3) | 1 (1)
Tremor (Nervous system disorders) | 3 (4) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrocalcinosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 4 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (6) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Link to the full study results: https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17902

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Depending on local requirements, Sponsor's consent necessary before publication of study, or Sponsor can review results communications before public release with a right to request changes to communications regarding trial results between 40 to 60 and up to 90 or 120 days, as applicable, from the time submitted to Sponsor for review to remove references to Sponsor's Confidential Information or delay results communications to permit Sponsor to obtain appropriate Intellectual Property protection.

DOCUMENTS (2):
  • Study Protocol (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT03505099/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT03505099/SAP_001.pdf